CLINICAL TRIAL: NCT04947475
Title: Project MATLINK: Development and Evaluation of a Screening, Brief Intervention, & Referral to Treatment (SBIRT) Program for Opioid Dependent Prisoners and Probationers Transitioning to the Community
Acronym: MATLINK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Ukrainian Institute on Public Health Policy (Other); AFEW Kyrgyzstan (Unknown); AFI - Act For Involvement (Unknown); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 1407014374; 2R01DA029910-06 (NIH)
Record Dates: First submitted 2021-06-23; First posted 2021-07-01 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Opioid-use Disorder; HIV Infections; Tuberculosis; Hepatitis C; Hepatitis B; Depression; Syphilis
Keywords: HIV; OUD; Methadone; HCV; HBV; TB; Depression; Syphilis
MeSH Terms: conditions — Opioid-Related Disorders; HIV Infections; Tuberculosis; Hepatitis C; Hepatitis B; Depression; Syphilis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Screening, Brief Intervention, & Referral to Treatment (SBIRT) Program (Experimental): There are two objectives to the Brief Intervention. First, the BI is designed to inform potential participants on the risks of substance misuse, abuse, and dependency by illustrating the potential hazards and adverse health consequences. Second, the BI aims to motivate potential participants to reduce risky behavior (e.g., continued drug use) and seek treatment for their substance dependence disorder.
  Interventions: Behavioral: SBIRT

INTERVENTIONS:
Behavioral: SBIRT — First, the BI is designed to inform potential participants on the risks of substance misuse, abuse, and dependency by illustrating the potential hazards and adverse health consequences. Second, the BI aims to motivate potential participants to reduce risky behavior (e.g., continued drug use) and seek treatment for their substance dependence disorder. In our BI, we will provide evidence-based information on Opioid Agonist Therapy (OAT) that is available to them in the community upon release or in the community. We will inform them of the risks and benefits of OAT and explain to them how OAT can be accessed in the community. OAT is provided at no cost to Ukrainian, Moldovan, and Kyrgyz citizens with opioid dependence. The BI will last approximately 20 minutes and time will be made available for them to ask questions. The BI will not be audio recorded.

SUMMARY:
The purpose of this study is to evaluate the efficacy a Screening, Brief Intervention, and Referral to Treatment (SBIRT) program for linking opioid dependent individuals currently incarcerated or in probation in Moldova, Kyrgyzstan, and Ukraine to opioid substitution therapy in the community after release or during their probation period.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. Within 180 days of release or possible release (eligible for parole) to the community, but greater than 7 days to release to the community OR currently in probation.
3. FOR THOSE IN PRISON: Relocating to a location within 30 km (approximately 60-minute commute) of the referred Narcology center. Each participant will be asked the address he/she is planning to reside under that will be immediately checked on the map to determine the travel time. A participant then will be asked if he/she would be willing to travel the distance to a particular OAT site. If a person does not meet this inclusion criterion, he/she will be referred to a local harm reduction center.
4. Meets ICD-10 screening criteria for pre-incarceration opioid dependence

   FOR THOSE IN PROBATION:
5. Living within 30 km of an OAT delivery site
6. Not having received OAT in the last 15 days.
7. Positive for OUD

Exclusion Criteria:

1. Pregnant or may become pregnant
2. FOR THOSE IN PRISON: Will be released from prison in 7 days or less.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 835 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Enrollment on OAT | 12 months
  Total number of participants who enroll on OAT divided by the number of participants who underwent study procedures, per country.

SECONDARY OUTCOMES:
OAT Knowledge | 6 month
  Overall mean change in composite score of knowledge of OAT pre vs post intervention stratified by study groups (enrolled vs not en rolled on OAT) at the 6-month mark.
OAT Attitudes | 6 months
  Overall mean change in composite score of attitudes towards OAT pre vs post intervention stratified by study groups (enrolled vs not en rolled on OAT) at the 6-month mark.
Interest in OAT | 6 months
  Overall mean change in composite score of interest in initiating OAT pre vs post intervention stratified by study groups (enrolled vs not en rolled on OAT) at the 6-month mark.
OAT Difficulty | 6 months
  Overall mean change in composite score of difficulty in initiating OAT pre vs post intervention stratified by study groups (enrolled vs not en rolled on OAT) at the 6-month mark.
OAT Importance | 6 months
  Overall mean change in composite score of importance of initiating OAT pre vs post intervention stratified by study groups (enrolled vs not en rolled on OAT) at the 6-month mark.

CONTACTS AND LOCATIONS:
Overall Officials: Frederick L Altice, MD, Principal Investigator — Yale University; Natalya Shumskaya, Study Director — AIDS Foundation East-West; Nataliia Saishuk, Study Director — Ukrainian Institute for Public Health Policy; Svetlana Doltu, Study Director — AFI - Act For Involvement
Locations (3):
- AIDS Foundation East-West, Bishkek, Kyrgyzstan
- AFI - Act for Involvement, Chisinau, Moldova
- Ukrainian Institute for Public Health Policy, Kyiv, Ukraine

IPD SHARING:
Plan to Share IPD: Undecided